CLINICAL TRIAL: NCT05764603
Title: Comparison of Conventional MRI,MR Arthrography and MSCT Arthrography in the Detection and Grading of Chondral Lesions of the Osteo Arthritic Knee
Brief Title: Comparison Between MR Arthrography ,ct Arthrography and Conventional MR in Osteoachondral Lesions of Knee Osteo Arthritis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Bakheet, doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 04-2023-100016
Record Dates: First submitted 2023-01-23; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: mri and ct arthrography
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental)
  Interventions: Drug: MRI

INTERVENTIONS:
Drug: MRI — MR ARTHROGRAPHY AND CT ARTHROGRAPHY IN PATIENT WITH KNEE OSTEOARTHRITIS
  Other Names: CT

SUMMARY:
The aim of this study is to compare the diagnostic efficacy of conventional MRI, MR arthrography and MDCT arthrography in the detection and grading of chondral lesions of the osteoarthritic knee with arthroscopic correlation

DETAILED DESCRIPTION:
The knee is a diarthrodial joint formed by two joint surfaces: the tibiofemoral and patellofemoral surfaces. The medial and lateral tibiofemoral compartments, together with the patellofemoral joint, form the three compartment of the knee, and these are covered by hyaline articular cartilage. Hyaline articular cartilage is a kind of dense conjunctive tissue consisting of cells, water and matrix. The normal hyaline cartilage is well-structured and elastic, with a smooth surface and its functions to protect the subchondral bone, allow the articular surfaces to slide across each other without friction and absorb impact. Damage of the articular cartilage is considered to be the hallmark of osteoarthritis (OA), even if other factors are involved in the pathogenesis of the disease (1). Knee osteoarthritis (OA) is a common progressive multifactorial joint disease and is characterized by chronic pain and functional disability. Knee OA accounts for almost four fifths of the burden of OA worldwide and increases with obesity and age (2). Knee osteoarthritis (OA) is often initially evaluated by plain x ray (AP, LAT) views which its useful technique for early diagnosis of OA whoever it is still limited imaging tool for detection of more findings as the disease progress including articular cartilage defect. Ultrasound is extremely sensitive for identifying synovial cysts that sometimes form in people with osteoarthritis. Ultrasound is excellent for evaluating the ligaments and tendons around the joint, which can be stretched or torn because of osteoarthritis and other advantages of ultrasound include its easy availability and multiplanar capability, as well as economic advantages but it has multiple disadvantages including that it is not suitable for evaluation the progression of OA (3). Magnetic resonance imaging (MRI) can provide the most comprehensive assessment of OA with the advantages of being noninvasive and multiplanar with excellent soft tissue contrast. However, MRI is expensive, time consuming, and not widely used for monitoring OA clinically. (3) MSCT can also be used to evaluate OA as can get an isotropic sub-millimeter spatial resolution with improved longitudinal resolution, The examination time is substantially reduced with decreased motion artifact, The cost is relatively lower than MRA in most countries(4) ,also useful in providing guidance for therapeutic and diagnostic procedure, even patients with metallic devices or implants, who are poorly indicated for MRA, can undergo the procedure, and we can easily estimate the lesion in the vicinity of metal without artifacts , but CTA may have some limitations in the evaluation of soft tissues and these are also invasive and require radiation exposure.(5) Magnetic resonance arthrography (MRA) and multi slice CT arthrography (MSCTA) of the knee are considered the best-performing imaging techniques in diagnosing knee osteo arthritis if prospectively compared with arthroscopic findings. These two imaging procedures are definitely better than plain CT or MRI of the knee because of the contrast resolution due to the presence of intraarticular diluted paramagnetic contrast or iodinated agent, respectively, and to the distension of the joint capsule. The evaluation of site, type, grade, and extent of the disease is more reliable. The two techniques give different information due to a higher CT sensitivity for calcifications and bone injuries and an optimal MR contrast resolution for soft tissue abnormalities (3) The combined use of iodinated contrast material for fluoroscopic confirmation of the articular position of the needle before injection of gadolinium chelates for MR arthrography offers the unique opportunity to compare CTA and MRA findings in carefully selected cases(6) Gadopentetate dimeglumine and iodinated contrast material can be mixed before MR imaging without any release of free gadolinium and are therefore safe for confirming the intraarticular placement of contrast material before MR arthrography (6)

ELIGIBILITY:
Inclusion Criteria:

* In this study 50 patients confirmed by X-ray to have early or advanced osteoarthritic changes which referred from the orthopedic clinic will be included

Exclusion Criteria:

* The exclusion criteria include fractures, septic knee, previous knee arthroscopy or open surgery. All metallic (non titanium) body implants that may include cardiac pacemakers, brain aneurysm clips, cochlear implants, vascular stents are considered an absolute contraindication to the performance of the procedure. Pregnancy (especially early pregnancy) is an absolute contraindication to the performance of MDCT (radiation exposure). Young patients below 18 years old..

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of conventional MRI, MR arthrography in diagnosis and grading of chondral lesions of the osteoarthritic knee | two years
  compare the MRI and MR arthrography in diagnosis and grading of severity of osteochondral lesions in knee osteoarthritis using I- V staging system
Comparison of conventional MRI, MSCT arthrography in diagnosis and grading of chondral lesions of the osteoarthritic knee | Two years
  compare the MRI and MSCT arthrography in diagnosis and grading of severity of osteochondral lesions in knee osteoarthritis using I- V staging system

REFERENCES:
- [Background] da Cunha Cavalcanti FM, Doca D, Cohen M, Ferretti M. UPDATING ON DIAGNOSIS AND TREATMENT OF CHONDRAL LESION OF THE KNEE. Rev Bras Ortop. 2015 Nov 16;47(1):12-20. doi: 10.1016/S2255-4971(15)30339-6. eCollection 2012 Jan-Feb. PMID 27027078
- [Background] Hunter DJ, Bierma-Zeinstra S. Osteoarthritis. Lancet. 2019 Apr 27;393(10182):1745-1759. doi: 10.1016/S0140-6736(19)30417-9. PMID 31034380
- [Background] Li Q, Amano K, Link TM, Ma CB. Advanced Imaging in Osteoarthritis. Sports Health. 2016 Sep;8(5):418-28. doi: 10.1177/1941738116663922. Epub 2016 Aug 10. PMID 27510507